CLINICAL TRIAL: NCT04800679
Title: Combination Therapy for PDR
Brief Title: Intravitreal Bevacizumab vs Laser vs Combination of Bevacizumab and Modified Laser in PDR
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Zahra Rabbani Khah, Head of ophthalmic research center, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 97378
Record Dates: First submitted 2019-12-28; First posted 2021-03-16 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2020-12

CONDITIONS: Proliferative Diabetic Retinopathy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- intravitreal bevacizumab injections and then rescue (Active Comparator)
  Interventions: Drug: receive 4 monthly IVB injections and then rescue IVB
- PRP group (Active Comparator)
  Interventions: Drug: PRP group
- IVB injections and a modified laser (Active Comparator)
  Interventions: Drug: IVB injections and a modified laser

INTERVENTIONS:
Drug: receive 4 monthly IVB injections and then rescue IVB — IVB group that receive 4 monthly IVB injections and then rescue IVB
  Arms: intravitreal bevacizumab injections and then rescue
Drug: PRP group — PRP group that undergo full PRP in 2 or 3 sessions and then rescue IVB
  Arms: PRP group
Drug: IVB injections and a modified laser — Combination group that receive 2 bimonthly IVB injections and a modified laser (1 session anterior to the equator) and then rescue IVB or laser
  Arms: IVB injections and a modified laser

SUMMARY:
In this randomized 3-armed clinical trial, 105 eyes with PDR will be included and divided randomly into 3 groups: IVB group (35 eyes) that receive 4 monthly IVB injections and then rescue IVB, PRP group (35 eyes) that undergo full PRP in 2 or 3 sessions and then rescue IVB, and combination group (35 eyes) that receive 2 bimonthly IVB injections and a modified laser (1 session anterior to the equator) and then rescue IVB or laser. Diabetic macular edema (DME) will be treated independently in all groups by IVB. Primary outcome will be the number and activity of neovascularizations at 4,8 and 12 months and secondary measures will be changes in best corrected visual acuity (BCVA) and central macular thickness (CMT), and number of examinations and injection.

ELIGIBILITY:
Inclusion Criteria:

* Presence of PDR with the indication of full PRP according the intend of investigator
* Best corrected visual acuity of 20/320 or better
* Media clarity, pupillary dilation and patient's cooperation sufficient for full PRP, wide-field FAG and OCT

Exclusion Criteria:

* History of prior PRP with more than 100 burns outside the posterior pole
* Tractional retinal detachment involving the macula
* Evidence of neoplasia of angle on examination
* Macular edema due to a cause other than DME
* Any ocular condition which may change visual acuity during the study
* Substantial cataract which has declined the vision by 3 lines or more
* History of intravitreal injection of anti-VEGF agent in past 2 months
* History of any use of corticosteroid during past 4 months
* History of major intra-ocular surgery except cataract surgery
* History of YAG laser capsulotomy during past 2 months
* Aphakia and uncontrolled glaucoma according to investigator judgment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Extent of neovascular tissues in disc-diameter measured by investigator according to the wide-field FAG | 12 months
  Number of neovascular tissue counted by investigator according to FAG

SECONDARY OUTCOMES:
Best corrected visual acuity based on Snellen chart | 12 months
Central retinal thickness according to macular OCT | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Ophthalmic Research Center, Tehran, Iran

REFERENCES:
- [Derived] Shahraki T, Arabi A, Nourinia R, Beheshtizadeh NF, Entezari M, Nikkhah H, Karimi S, Ramezani A. PANRETINAL PHOTOCOAGULATION VERSUS INTRAVITREAL BEVACIZUMAB VERSUS A PROPOSED MODIFIED COMBINATION THERAPY FOR TREATMENT OF PROLIFERATIVE DIABETIC RETINOPATHY: A Randomized Three-Arm Clinical Trial (CTPDR Study). Retina. 2022 Jun 1;42(6):1065-1076. doi: 10.1097/IAE.0000000000003450. PMID 35594075